CLINICAL TRIAL: NCT03319992
Title: Robotic Assisted Task-Oriented Rehabilitation of Upper Limb for Chronic Stroke Patients
Brief Title: Upper Limb Task-Oriented Rehabilitation With Robotic Exoskeleton for Hemiparetic Stroke Patients
Acronym: RH-LEXOS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Scuola Superiore Sant'Anna di Pisa (Other)
Collaborators: Azienda Ospedaliero, Universitaria Pisana (Other)
Responsible Party: Principal Investigator, Antonio Frisoli, Prof, Office of Research and Development, Scuola Superiore Sant'Anna di Pisa
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RH-UL-LEXOS-10
Record Dates: First submitted 2017-10-20; First posted 2017-10-24 (Actual); Last update posted 2021-04-13 (Actual); Status verified 2021-04

CONDITIONS: Cerebrovascular Accident (CVA); Chronic Disease; Stroke Rehabilitation
Keywords: Robotics [H01.671.293.643]; Exoskeleton Device [E07.341]; Rehabilitation Research [H01.770.644.145.472]; Physical and Rehabilitation Medicine [H02.403.680]; Exercise Therapy [E02.779.483]; Patient Outcome Assessment [N05.715.360.575.575.399]
MeSH Terms: conditions — Stroke; Chronic Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional treatment (No Intervention): The conventional treatment arm was conducted according to a set of exercises that were specifically designed in order to match the robotic treatment. Patients received both physical therapy (PT) and occupational therapy (OT) session, administered by the physiotherapists of the hospital. The therapist will provide a specific conventional treatment comparable with the robotic treatment in terms of session time and therapeutic goals.
- Robotic treatment (Experimental): The patients enrolled in the robotic arm are going to be undergone a series of passive, assisted and active mobilization in upper limb task-oriented exercises implemented in 3d virtual environments. Briefly speaking, these tasks promote the upper arm multi-joints coordination during the execution of reaching movements and grasping actions of fixed virtual objects displaced in the space.
  Interventions: Device: Upper Arm Rehabilitation Light Exoskeleton (RH-LEXOS)

INTERVENTIONS:
Device: Upper Arm Rehabilitation Light Exoskeleton (RH-LEXOS) — RH-LEXOS is a robotic exoskeleton device to support the rehabilitation of stroke patients. This system is conceived for the force assistance, integrated in a Virtual Reality system that allows implementing rehabilitative exercises highly interactive and engaging for the patients. Passive, assisted and active mobilization of upper arm is provided through the use of the exoskeleton robotic device within high intensive, repetitive, task-oriented exercises and an objective and reliable mean for monitoring patients' progress.
  Arms: Robotic treatment

SUMMARY:
The aim of this study is to evaluate the effects of an assisted rehabilitation treatment through a robotic exoskeleton device on the functional recovery in a group of patients with hemiparesis from lesion of the first motor neuron (post-stroke), compared with a group of patients subjected to a conventional rehabilitation treatment. The patients enrolled in the study are chronic stroke injured with right hemiparesis of moderate to severe degree, by the system injury pyramid, never undergoing rehabilitation treatment with robots.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of a first-ever left hemisphere ischemic or hemorrhagic stroke at least 6 months prior to entry into the study;
* minimum ability for shoulder humeral elevation;
* upper-extremity motor function Fugl-Meyer (FM) score ≥ 15(out of 66);
* absence of neurological or muscular disorders that interfere with neuromuscular function;
* absence of severe cognitive deficits that would limit patients' ability to complete the study;
* minimum score of 2 in the Modified Ashworth Scale;
* not participating in any experimental rehabilitation or drug studies at the same time
* no previous experience with robotic treatments.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2016-07-20 (Actual); Primary Completion 2018-10-20 (Actual); Study Completion 2018-11-30 (Actual)

PRIMARY OUTCOMES:
Change in Fugl-Meyer Assessment (FMA( Score | baseline and 6 weeks
  The null hypothesis tested in this study was the change in motor function domain of the upper extremity portion of the Fugl-Meyer assessment in the Robotic Group (Robotic Treatment) would be the same as the one obtained by the Control Group (Conventional Treatment).
  The FMA outcome is further divided and analyzed in terms of sub-items. In particular, the motor FMA score is divided into proximal (shoulder and elbow movement, 36 points) and distal (hand and wrist movement, 24 points) sub-items.

SECONDARY OUTCOMES:
Functional scale: Bimanual Activity Test (BAT) | baseline and 6 weeks
  The BAT is a functional scale designed to quantify the contribution of patient's affected upper limb to execute 25 common Activities of Daily Living such as Loosen and tighten the cap of a bottle , or unscrew a bolt. The elapsed time for accomplishing each task is measured and the therapist also give a score (ranging from 1 to 4) about the quality of each movement.
  The BAT data is analyzed also in terms of sub-items, divided into pinch-tasks and power-tasks collecting those items requiring fine and gross manipulation motor skills respectively.
Modified Ashworth (MA) scale | baseline and 6 weeks
  The MA scale (Bohannon and Smith, 1987) is used to evaluate spasticity of the upper limb and to assess abnormal muscle tone at the shoulder and elbow. The MA scale is a 6-point scale: scores range from 0 to 4, where lower scores represent normal muscle tone and higher scores represent spasticity or increased resistance to passive movement. MA scores were averaged across the two joints and across testing directions (flexion, extension) to estimate abnormal muscle tone in the upper extremity (Zackowski, Dromerick et al., 2004)
Robotic kinesiological assessment of movement: Execution Time | At end of each session, during 6 weeks of enrollment in treatment
  This measure is evaluated only in the group of patients performing robotic training, at the end of each session through the analysis of their performance during the execution of an evaluation exercise without robotic assistance.The patients are instructed to reach different targets positioned in front of them and placed around a vertical circumference at 12 equally spaced locations.
  The robotic measure is extracted for each outgoing (from the center to the target) movement. The execution time is measured as the elapsed time (measure in seconds) for accomplishing each movement, measured from the time of grasping of the virtual object at the start position to the release time at the target position.
Robotic kinesiological assessment of movement: Smoothness index | At end of each session, during 6 weeks of enrollment in treatment
  This measure is evaluated only in the group of patients performing robotic training, at the end of each session through the analysis of their performance during the execution of an evaluation exercise without robotic assistance.The patients are instructed to reach different targets positioned in front of them and placed around a vertical circumference at 12 equally spaced locations.
  The robotic measure is extracted for each outgoing (from the center to the target) movement.
  The smoothness index is computed in the same interval period by counting the number of peaks in the velocity profile of movement, namely the Number of Movements Units (NMU) (Fasoli S, Krebs J Neurosci 2002)

CONTACTS AND LOCATIONS:
Overall Officials: Carmelo Carmelo, Carmelo, Study Director — U.O. Neurorehabilitation Division, Azienda Ospedaliero-Universitaria Pisana (AOUP)
Locations (1):
- University Hospital of Pisa, Pisa, Italy

IPD SHARING:
Plan to Share IPD: Undecided
De-identified individual participant data for all primary and secondary outcome measures will be made available

REFERENCES:
- [Derived] Frisoli A, Barsotti M, Sotgiu E, Lamola G, Procopio C, Chisari C. A randomized clinical control study on the efficacy of three-dimensional upper limb robotic exoskeleton training in chronic stroke. J Neuroeng Rehabil. 2022 Feb 4;19(1):14. doi: 10.1186/s12984-022-00991-y. PMID 35120546